CLINICAL TRIAL: NCT06629363
Title: Determinants of Malignant Hypertension Onset and Related Target Organ Damages: the HAMA Biobank
Acronym: HAMABANK
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier de PAU (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-A01738-41
Record Dates: First submitted 2024-10-01; First posted 2024-10-08 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Malignant Hypertension
Keywords: Malignant hypertension; severe hypertension; hypertensive emergency; target organ damage; pathophysiology; biomarkers
MeSH Terms: conditions — Hypertension, Malignant; Hypertension; Hypertensive Crisis | interventions — Biological Specimen Banks

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample for DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: biobank — The following samples will be collected :
  * Serum samples and plasma sample: inclusion visit and follow up visit
  * Urines samples : inclusion visit and follow up visit
  * blood DNA: inclusion visit
  * Blood RNA: inclusion visit and follow up visit

SUMMARY:
The HAMA bank is an initiative aimed at collecting, preparing, and storing biological samples from patients treated for malignant hypertension and included in the HAMA cohort. Conducted under CRB (ISO20387) conditions, this biobank serves as an essential resource for understanding the disease's pathophysiology, as well as for identifying novel biomarkers and therapeutic targets

DETAILED DESCRIPTION:
Malignant hypertension (MH) is an acute and severe form of hypertension that can lead to rapid target organ damage and potentially be fatal within months if not treated. Despite the severity, MH manifests in various phenotypes, suggesting multiple underlying pathophysiological pathways. The HAMA bank aims to address this by collecting biological samples at two distinct time-points:

For " Pre-existing Patients " in the HAMA cohort: A one-time collection focused on genetic analysis. A full sample (equivalent to sample 1 below) may be collected in option.

For Newly Diagnosed Patients (Incident Patients): Sample 1 "Acute Phase": Collected between Day 0 and Day 7 post-admission to any HAMA recruiting centers. This will be used for initial multi-omics analysis. Sample 2 "Chronic Phase": Collected between the 1st and 6th months during a follow-up visit at the investigating center.

These samples will be cross-referenced with clinical and biological data from the HAMA cohort. The cohort follow-up schedule is: 1, 3, 6, 12 months after MH diagnosis and annually for a total of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* patients included in the HAMA cohort with the following critera :

  * Malignant hypertension according to the classic definition (Severe hypertension associated with severe hypertensive retinopathy)
  * Severe hypertension associated with acute target organ damage due to high blood pressure

Exclusion Criteria:

* Refusal to participate to the substudy " HAMA bank "
* patient on chronic dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with malignant hypertension
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2036-04-01 (Estimated); Study Completion 2036-04-01 (Estimated)

PRIMARY OUTCOMES:
Decipher the mechanisms responsible for the transition from severe to malignant hypertension | At inclusion and 6 month
  Compare the multiomic signature of patients admitted for malignant hypertension, between MHT acute crisis (admission) and resolution (6 month later). Transcriptomic, proteomic and metabolomic evolution between these 2 time points and focus on genetic background in relevant system, like angiogenic, vasoactif system, complement system and inflammasome will be described.

SECONDARY OUTCOMES:
Understand the determinants of the heterogeneity in target organs damages (TOD) during MHT crisis | At inclusion
  Patient's multiomic signature according to the number of target organ damage presented by the patients, the presence and severity of each TOD (heart, brain, kidney, retina and endothelium) will be compared
Focus on the role of complement system in MHT crisis | At inclusion and 6 month
  level of circulating complement factors and transcripts between the admission (acute phase of malignant hypertension) and the follow-up consultation will be specificaly compared. Prevalence of pathogenic variant involved in the complement system in the study population will described.

CONTACTS AND LOCATIONS:
Overall Officials: Romain BOULESTREAU, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: Undecided